CLINICAL TRIAL: NCT02295059
Title: Omega-3 Fatty Acids and ERPR(-) and HER-2/Neu(+/-) Breast Cancer Prevention
Brief Title: Omega 3 Fatty Acids and ERPR(-)HER2(+/-) Breast Cancer Prevention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16421; 1R01CA164019-01A1 (NIH)
Record Dates: First submitted 2014-10-14; First posted 2014-11-20 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Breast cancer; ERPR negative; HER-2/neu overexpression positive or negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Fatty Acids, Omega-3; Fish Oils; Eicosapentaenoic Acid; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega 3 fatty acids - high dose (Experimental): ~5 g EPA+DHA in 5 capsules per day
  Interventions: Dietary Supplement: omega 3 fatty acids
- Omega 3 fatty acids - low dose (Experimental): ~0.9 g EPA+DHA + fatty acids based on the typical American diet in 5 capsules per day
  Interventions: Dietary Supplement: omega 3 fatty acids

INTERVENTIONS:
Dietary Supplement: omega 3 fatty acids — supplied as soft gelatin capsules for oral administration
  Other Names: fish oil; eicosapentaenoic acid; docosahexaenoic acid

SUMMARY:
The study aims to determine biological changes associated with a low vs high dose of omega 3 fatty acids, docosahexaenoic acid (DHA), eicosapentaenoic acid (EPA), over 12 months in women at risk for recurrent breast cancer. The objectives of the trial are to develop mammary epithelial, adipose tissue specific markers of exposure and response to omega 3 fatty acid supplements that can be carried forward into definitive intervention trials of omega 3 fatty acids for breast cancer prevention. The investigators will randomize 80 subjects with hormone receptor negative, HER-2/neu overexpression positive or negative breast cancer to either a high or low dose of omega 3 fatty acids. Using fine needle aspiration to procure cellular samples of breast epithelial and adipose tissue, the investigators will determine the effects of omega 3 fatty acids on mammary specific biomarkers of response.

DETAILED DESCRIPTION:
The study aims to determine biological changes that occur with a 12 month intervention of low (~0.9 g EPA+DHA/day) vs high dose (~5.4 g EPA+DHA/day) of omega 3 polyunsaturated fatty acids (PUFAs) in women survivors of hormone unresponsive breast cancer. The objectives of the trial are to develop unique mammary epithelial, adipose tissue specific markers of exposure and response to omega 3 fatty acid supplements that can be carried forward into definitive intervention trials of EPA, DHA/omega 3 PUFAs for breast cancer prevention. The investigators will randomize 80 subjects with hormone receptor negative, HER-2/neu overexpression positive or negative breast cancer to either a high or low dose of omega 3 PUFAs. Using fine needle aspiration to procure cellular samples of breast epithelial and adipose tissue, the investigators will determine the effects of omega 3 fatty acids on mammary specific biomarkers of response.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of Stage 0 to III breast cancer that is estrogen receptor negative, progesterone receptor negative with completion of definitive surgery, radiation therapy and/or chemotherapy.
* Completion of chemotherapy or trastuzumab for > six months and of radiation therapy for > 2 months, as applicable and 5 years or less from completion of standard therapy.
* Greater than 1 year from pregnancy, lactation.
* Mammogram within the eight months prior to study enrollment that is not suspicious for breast cancer (ACR Class I-III).

Exclusion Criteria:

* Other current malignancy or metastatic malignancy of any kind.
* Ongoing chemotherapy, radiation therapy, or other cancer-related treatment.
* Subjects on Coumadin or other anticoagulants.
* Subjects with breast implants.
* Subjects who have had radiation to both breasts or who have undergone bilateral mastectomies.
* Barriers to fine needle aspiration sampling of breast adipose tissue and/or parenchymal breast tissue, including breast implants, history of radiation to both breasts, bilateral mastectomies, and/or insufficient breast adipose/parenchymal tissue for adequate fine needle aspiration (FNA) sampling.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, hypertension, or psychiatric illness/social situation that would limit compliance with study requirements.
* Chronic use of omega 3 fatty acid concentrates or capsules within the 3 months prior to entry on the study or any other supplements that might interact with omega 3 fatty acid supplements.
* Pregnant or nursing women.
* Known sensitivity or allergy to fish.
* Subjects on a standing regimen of full dose aspirin (greater than 325 mg/day), NSAIDs (nonsteriodal anti inflammatory drug) or NSAID-containing products.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-08-09 (Actual); Primary Completion 2026-06-22 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Changes in eicosanoids/metabolites including PGE2, PGE3 in breast adipose tissue | Baseline to up to 12 months
  Biomarker

SECONDARY OUTCOMES:
Changes in cytomorphology and/or cell proliferation of mammary epithelial cells | Baseline to up to 12 months
  Biomarker
Changes in DNA promoter methylation and pro-inflammatory gene expression in mammary epithelial and adipose tissue | Baseline to up to 12 months
  Biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Lisa D Yee, MD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frankhouser DE, DeWees T, Snodgrass IF, Cole RM, Steck S, Thomas D, Kalu C, Belury MA, Clinton SK, Newman JW, Yee LD. Randomized dose-response trial of n-3 fatty acids in hormone receptor negative breast cancer survivors - impact on breast adipose oxylipin and DNA methylation patterns. Am J Clin Nutr. 2025 Jul;122(1):70-82. doi: 10.1016/j.ajcnut.2025.04.021. Epub 2025 Apr 25. PMID 40288580